CLINICAL TRIAL: NCT06652516
Title: Study of Centrifugal Therapeutic Plasma Exchange and Membrane Therapeutic Plasma Exchange; a Comparative Study
Brief Title: Comparison Between Centrifugation Based and Membrane Based Plasma Exchange
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB NO: 00012098
Record Dates: First submitted 2024-10-07; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Therapeutic Plasma Exchange
MeSH Terms: interventions — Plasma Exchange

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cTPE (Active Comparator): This group performed the first session of plasma exchange by centrifugation and the second session by membrane filtration
  Interventions: Procedure: plasma exchange
- mTPE (Active Comparator): This group performed the first session of plasma exchange by membrane filtration and the second session by centrifugation
  Interventions: Procedure: plasma exchange

INTERVENTIONS:
Procedure: plasma exchange — comparison between the 2 methods of plasma exchange as regards efficacy, performance and adverse events.
  Procedure of therapeutic plasma exchange (TPE) :
  mTPE will be done by bellco hemodialysis machine (Formula 2000), while cTPE will be done by Nigale Plasma Collector (XJC 2000). The vascular access used for both types of plasma exchange will be central venous catheter inserted into the internal jugular vein, subclavian or femoral vein.
  Prescription of TPE The amount of plasma to be treated is usually equivalent to the patient's estimated plasma volume (EPV).
  Estimated plasma volume will be calculated using the following formula (Kaplan formula) in litres:
  * EPV = 0.07 x wt (kg) x (1 - hematocrit) in males.
  * EPV = 0.065 x wt (kg) x (1 - hematocrit) in females.

SUMMARY:
This study aims at comparing centrifugation based therapeutic plasma exchange (cTPE) versus membrane based therapeutic plasma exchange (mTPE) as regards performance, effectiveness and adverse events in patients indicated for TPE.

DETAILED DESCRIPTION:
* Study setting: Patients of this study were recruited from the hemodialysis unit of Alexandria Main University Hospital.
* Study design: Randomized prospective crossover study.
* Study population: Twenty patients having clinical indication for TPE.
* They were divided into 2 groups by 1 to 1 randomization Group A: ten patients received the first session of TPE by cTPE and the second session was performed by mTPE 48 hours later.

Group B: ten patients received the first session of TPE by mTPE and the second session was performed by cTPE 48 hours later.

Only the results of 2 sessions for each group were recorded in the study, even if the patients needed further sessions of TPE.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged more than 18 years old having indication for plasma exchange (based on American Society for Apheresis (ASFA) therapeutic category 1, 2, 3).

  * Category I: includes disorders for which TPE is accepted as first-line therapy, either as primary stand-alone treatment or in conjunction with other modes of treatment. Examples include Guillain-Barre syndrome, acquired thrombotic thrombocytopenic purpura, and erythrocytapheresis in sickle cell diseases with certain complications (eg, stroke).
  * Category II: includes disorders for which TPE is accepted as second-line therapy, either as a stand-alone treatment or in conjunction with other modes of treatment. Examples include life-threatening hemolytic anemia for cold agglutinin disease or Lambert-Eaton myasthenic syndrome.
  * Category III: includes disorders for which the optimum role of apheresis therapy is not established. Decision making should be individualized. Examples include TPE for hyper-triglyceridemic pancreatitis or extracorporeal photopheresis for nephrogenic systemic fibrosis.
* Approval to sign a written consent.

Exclusion Criteria:

* Refusal to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Time to setup and prime the machine (in minutes) | immediately after plasma exchange procedure
Procedure time (in minutes). | immediately after plasma exchange procedure
Time to exchange 1 litre of plasma (in minutes). | immediately after plasma exchange procedure
Blood flow rate (ml/minutes) | immediately after plasma exchange procedure
Plasma removal efficiency (PRE). | immediately after plasma exchange procedure
  Plasma removal efficiency is an established metric used to analyse the performance of an apheresis device during a TPE procedure. It represents the fraction of plasma that has been removed in a TPE procedure in relation to the plasma that has been processed.
Efficacy in clearance of interleukin 6 and tumor necrosis factor alpha | immediately after plasma exchange procedure
  serum level of interleukin 6 and tumor necrosis factor apha were assessed before and after each session of therapeutic plasma exchange
Adverse events | immediately after plasma exchange procedure
  All adverse events occurring during the session were reported including any of the following
  * Hemolysis.
  * Urticaria.
  * Hypotension.
  * Hypocalcemia.
  * Clotting of the extracorporeal circuit.
  * Others.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham A Elghoneimy, MD, Principal Investigator — Department of internal medicine, nephrology unit, Alexandria faculty of medicine, Egypt
Locations (1):
- Alexandria university, Faculty of medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elghoneimy HA, Elkader MMA, Saad NLM, Tawfiq AA, El-Wakil HS. Study of Centrifugal Therapeutic Plasma Exchange and Membrane Therapeutic Plasma Exchange; A Comparative Study. Ther Apher Dial. 2025 Dec 21. doi: 10.1002/1744-9987.70104. Online ahead of print. PMID 41422826